CLINICAL TRIAL: NCT04584177
Title: Arm-hand Boost Program During Inpatient Rehabilitation After Stroke: Pilot Randomized Controlled Trial
Brief Title: Arm-hand Boost Program During Inpatient Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Study 19.27
Record Dates: First submitted 2020-09-04; First posted 2020-10-12 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm-hand BOOST + Control (Experimental): First 4 weeks arm-hand boost program, afterwards, 4 weeks of control program
  Interventions: Behavioral: Arm-hand BOOST program; Behavioral: Control program
- Control + Arm-hand BOOST (Experimental): First 4 weeks control program, afterwards 4 weeks arm-hand boost program
  Interventions: Behavioral: Arm-hand BOOST program; Behavioral: Control program

INTERVENTIONS:
Behavioral: Arm-hand BOOST program — The arm-hand boost program is provided 1 hour/day, 5x/week for 4 weeks, on top of their usual care program. The focus of the boost program is on scapula-setting, core-stability when reaching, movements with 30-60° flexion/abduction in shoulder, fine manipulation and integration in complex ADL tasks. Additionally, patients exercise 1 hour per week using the Armeo Power (Hocoma). Therefore, the additional arm-hand boost program consists of 24 one-hour sessions, provided over four weeks.
Behavioral: Control program — A dose-matched program of strengthening exercises for the lower limbs and general reconditioning

SUMMARY:
A pilot cross-over RCT including participants with sub-acute stroke is conducted in an inpatient rehabilitation setting. The experimental group (EG) receives an arm-hand boost program on top of their usual care program. The control group (CG) receives a dose-matched program of strengthening exercises for the lower limbs and general reconditioning. After 4 weeks, a cross-over is performed. Before, after 4 weeks and after 8 weeks of additional therapy, different clinical outcome measures for the upper limb are administered.

ELIGIBILITY:
Inclusion Criteria:

* first stroke, as defined by WHO,
* minimal stay of 4 weeks in inpatient setting at study start
* minimally 18 years old
* being able to sit independently (trunk control test, item 3 = 25),
* motor impairment in the upper limb (Fugl-Meyer assessment, stage 2 (synergies): 8-17p, or stage 2: <8p combined witht stage 5 (hand): >6p
* sufficient cooperation to perform intervention and evaluations

Exclusion Criteria:

* musculoskeletal and/or other neurological impairments with permanent damage that may hinder the study
* subdural hematoma, tumor, encephalitis, trauma, or other that lead to similar symptoms as stroke
* severe communication, cognitive or language impairments that hinder the investigations
* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Change from Fugl-Meyer Assessment-Upper Extremity at 4 weeks | Between baseline and first 4 weeks of study
  UL assessment - Function
Change from Fugl-Meyer Assessment-Upper Extremity at 8 weeks | Between baseline and end of study (=8 weeks)
  UL assessment - Function
Change from Action Research Arm Test at 4 weeks | Between baseline and first 4 weeks of study
  UL Assessment - Activities
Change from Action Research Arm Test at 8 weeks | Between baseline and end of study (=8 weeks)
  UL Assessment - Activities

SECONDARY OUTCOMES:
Change from Jebsen Taylor hand function test at 4 weeks | Between baseline and first 4 weeks of study
  UL Assessment - Activities
Change from Jebsen Taylor hand function test at 8 weeks | Between baseline and end of study (=8 weeks)
  UL Assessment - Activities
Change from Rivermead Motor Assessment Arm function at 4 weeks | Between baseline and first 4 weeks of study
  UL Assessment - Activities
Change from Rivermead Motor Assessment Arm function at 8 weeks | Between baseline and end of study (=8 weeks)
  UL Assessment - Activities
Change from Stroke upper limb capacity scale (SULCS) at 4 weeks | Between baseline and first 4 weeks of study
  UL Assessment - Activities
Change from Stroke upper limb capacity scale (SULCS) at 8 weeks | Between baseline and end of study (=8 weeks)
  UL Assessment - Activities
Change from Box & Block test at 4 weeks | Between baseline and first 4 weeks of study
  UL Assessment - Activities
Change from Box & Block test at 8 weeks | Between baseline and end of study (=8 weeks)
  UL Assessment - Activities

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Meyer, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Campus Sint-Ursula, Herk-de-Stad, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer S, Verheyden G, Kempeneers K, Michielsen M. Arm-Hand Boost Therapy During Inpatient Stroke Rehabilitation: A Pilot Randomized Controlled Trial. Front Neurol. 2021 Feb 26;12:652042. doi: 10.3389/fneur.2021.652042. eCollection 2021. PMID 33716948